CLINICAL TRIAL: NCT04951726
Title: Evaluating the Safety and Efficacy of Different Routes of Neostigmine Administration for Acute Colonic Pseudo Obstruction: a Prospective Randomized Trial
Brief Title: Neostigmine Route for Acute Colonic Pseudo Obstruction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Meghan Lewis, Assistant Professor of Clinical Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-07318
Record Dates: First submitted 2021-05-05; First posted 2021-07-07 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Ogilvie Syndrome
MeSH Terms: conditions — Colonic Pseudo-Obstruction | interventions — Neostigmine

STUDY DESIGN:
Intervention Model Description: Prospective randomized non-inferiority trial 2 Arms:
  1. 1.0 mg subcutaneous repeated q8hr until resolution for up to 24 hours (3.0 mg total in 24 hours)
  2. 2 mg slow intravenous injection over five minutes repeated q6hr until resolution for up to 24 hours. (8 mg total in 24 hours) (CONTROL GROUP)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IV push (Active Comparator): 2 mg slow intravenous injection over five minutes repeated q12hr until resolution for up to 24 hours. (4 mg total in 24 hours)
  Interventions: Drug: Neostigmine
- subcutaneous (Experimental): 1.0 mg subcutaneous repeated q8hr until resolution for up to 24 hours (3.0 mg total in 24 hours)
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Neostigmine — cholinesterase inhibitor
  Other Names: Bloxierz; Vagostigmin; Prostigmin

SUMMARY:
Neostigmine is commonly used for medical treatment of acute colonic pseudo obstruction, however, the ideal route of administration has not been determined. Though IV push works rapidly, it is likely associated with the most side effects. This study will compare the efficacy and side effect profile of 2 potential routes of administration: IV push and subcutaneous.

DETAILED DESCRIPTION:
Acute colonic pseudo-obstruction (ACPO) is a severe form of colonic ileus seen in patients hospitalized with a variety of medical and surgical conditions. The most serious complication is spontaneous colonic perforation, which occurs in 3% of cases with a mortality rate of up to 50%. The risk of perforation is greater in those patients with a cecal diameter >12 cm, although the duration of dilation might be more important than the cecal diameter. A significant number of patients will respond to the conservative measures enumerated in the abstract.

Endoscopic decompression of the dilated colon is undertaken commonly to prevent spontaneous perforation. However, it is performed under suboptimal conditions (unprepared and distended colon) increasing the risk of complications with a morbidity rate of 3% and a mortality rate of 1%. Furthermore, although effective initially in 69% of cases, 40% of them will have at least one recurrence. To decrease this recurrence rate, endoscopic placement of a drainage tube is now advocated. Patients who fail to respond to conservative therapy and colonoscopic decompression will require surgery, which has a mortality rate of up to 26%.

In an effort to find a more effective, noninvasive therapy, Ponec et al., introduced and highlighted the effect of IV neostigmine (2 mg over 3-5 min). Neostigmine was significantly more effective than placebo in rapidly decreasing colonic dilation in the majority of patients with ACPO. Although it has a short half-life, a single IV dose of 2 mg of neostigmine was sufficient in most cases to restore colonic motility.

It is important to be aware of contraindications to using parasympathetic agents, including bradyarrhythmia and history of bronchospasm. Patients need to be monitored while neostigmine is infused, and atropine should be available in the event of complications. Patients with renal insufficiency might be at higher risk of complications as a significant quantity of the drug is excreted in urine.

In light of these contraindications, administration by the subcutaneous (SQ) route has been utilized intermittently for ACPO. Data for use of SQ administration of neostigmine in adult patients are limited to one multi-institutional observational study, one case series, and two case reports in acute medical and palliative care patients. Although these case reports describe a range of dosing, the SQ route of administration appears to be attractive alternative to IV administration for this indication, with a time to effect of 8 to 10 hours.

This study is a prospective randomized non-inferiority trial that seeks to analyze the success of two different routes of neostigmine administration, sub-cutaneous and IV push, for safety and efficacy in the ACPO patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with radiologically confirmed acute colonic pseudo obstruction (ACPO).

   1. Plain abdominal radiograph or computed tomography imaging
   2. Cecal diameter of >9 cm or transverse colon diameter of >6 cm
2. Distal obstruction ruled out on imaging (Contrast enema, endoscopy, CT scan)

Exclusion Criteria:

1. Patients with previous neostigmine administration during current hospitalization
2. Patients with prior attempt at endoscopic decompression on this admission.
3. Patients with base-line heart rate of less than 60 beats per minute or on beta blocker medication
4. Patients with systolic blood pressure of less than 90 mm Hg
5. Signs of bowel perforation, with peritoneal signs on physical examination or free air on radiographs
6. Active bronchospasm requiring medication
7. Treatment with prokinetic drugs such as cisapride or metoclopramide in the 24 hours before evaluation
8. A history of colon cancer or partial colonic resection
9. Signs concerning for colonic obstruction
10. Active gastrointestinal bleeding
11. Pregnancy
12. Serum creatinine concentration of more than 3 mg per deciliter (265μmol per liter).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with radiographic resolution of colonic pseudo obstruction | 24 hours
  Number of patients who have cecal diameter <9 cm AND transverse diameter <6 cm on abdominal x-ray within 24h of initiation of neostigmine therapy.

SECONDARY OUTCOMES:
Number of patients with recurrence of colonic pseudo obstruction | 7 days
  Number of patients with recurrence of cecal diameter >9cm or transverse colon diameter >6cm
Number of patients with adverse medication reactions | 24 hours
  Number of patients that experience cardiac arrest; bradycardia, defined as a heart rate less than 60 beats/min; sustained hypotension, defined as a mean arterial pressure (MAP) less than 60 >2 min, bronchospasm documented in the medical record and needing emergent administration of albuterol or ipratropium-albuterol within 30 minutes of the dose; nausea documented in the medical record and need for emergent administration of an antiemetic within 30 minutes of the dose; or severe salivation, lacrimation, or diarrhea leading to drug discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Lewis, MD, Principal Investigator — University of Southern California
Locations (1):
- Los Angeles University of Southern California Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeMets DL, Lan KK. Interim analysis: the alpha spending function approach. Stat Med. 1994 Jul 15-30;13(13-14):1341-52; discussion 1353-6. doi: 10.1002/sim.4780131308. PMID 7973215
- [Background] Frankel A, Gillespie C, Lu CT, Hewett P, Wattchow D. Subcutaneous neostigmine appears safe and effective for acute colonic pseudo-obstruction (Ogilvie's syndrome). ANZ J Surg. 2019 Jun;89(6):700-705. doi: 10.1111/ans.15265. Epub 2019 May 13. PMID 31083785
- [Background] Ponec RJ, Saunders MD, Kimmey MB. Neostigmine for the treatment of acute colonic pseudo-obstruction. N Engl J Med. 1999 Jul 15;341(3):137-41. doi: 10.1056/NEJM199907153410301. PMID 10403850
- [Background] Kram B, Greenland M, Grant M, Campbell ME, Wells C, Sommer C. Efficacy and Safety of Subcutaneous Neostigmine for Ileus, Acute Colonic Pseudo-obstruction, or Refractory Constipation. Ann Pharmacother. 2018 Jun;52(6):505-512. doi: 10.1177/1060028018754302. Epub 2018 Jan 23. PMID 29359574
- [Background] Ilban O, Cicekci F, Celik JB, Bas MA, Duman A. Neostigmine treatment protocols applied in acute colonic pseudo-obstruction disease: A retrospective comparative study. Turk J Gastroenterol. 2019 Mar;30(3):228-233. doi: 10.5152/tjg.2018.18193. PMID 30541715
- [Background] van der Spoel JI, Oudemans-van Straaten HM, Stoutenbeek CP, Bosman RJ, Zandstra DF. Neostigmine resolves critical illness-related colonic ileus in intensive care patients with multiple organ failure--a prospective, double-blind, placebo-controlled trial. Intensive Care Med. 2001 May;27(5):822-7. doi: 10.1007/s001340100926. PMID 11430537
- [Background] Sgouros SN, Vlachogiannakos J, Vassiliadis K, Bergele C, Stefanidis G, Nastos H, Avgerinos A, Mantides A. Effect of polyethylene glycol electrolyte balanced solution on patients with acute colonic pseudo obstruction after resolution of colonic dilation: a prospective, randomised, placebo controlled trial. Gut. 2006 May;55(5):638-42. doi: 10.1136/gut.2005.082099. Epub 2005 Nov 23. PMID 16306137
- [Background] Vogel JD, Feingold DL, Stewart DB, Turner JS, Boutros M, Chun J, Steele SR. Clinical Practice Guidelines for Colon Volvulus and Acute Colonic Pseudo-Obstruction. Dis Colon Rectum. 2016 Jul;59(7):589-600. doi: 10.1097/DCR.0000000000000602. No abstract available. PMID 27270510